CLINICAL TRIAL: NCT03766867
Title: Interventional, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Initial Administration of 25 mg Vortioxetine Intravenously With 10 mg/Day Vortioxetine Orally in Patients With Major Depressive Disorder
Brief Title: Vortioxetine Intravenous Infusion at Initiation of Oral Treatment With Vortioxetine in Patients With Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17915A
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine infusion 25 mg; Drug: Vortioxetine tablets 10 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo infusion; Drug: Placebo tablets

INTERVENTIONS:
Drug: Vortioxetine infusion 25 mg — 1 mg/mL, concentrate for solution for infusion, 25 mL (25 mg) administered in 250 mL saline over 2 hours as single dose for 7 days
  Arms: Vortioxetine
Drug: Vortioxetine tablets 10 mg/day — 10 mg, tablets, oral administration once daily
  Other Names: Brintellix ®
  Arms: Vortioxetine
Drug: Placebo infusion — concentrate for solution for infusion, 25 mL administered in 250 mL saline over 2 hours as single dose
  Arms: Placebo
Drug: Placebo tablets — oral administration once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vortioxetine given as a single intravenous dose of 25 mg at initiation of an oral vortioxetine regimen of 10 mg/day for 7 days

DETAILED DESCRIPTION:
The study consists of a 7-day double-blind Treatment Period (Day 0 to Day 6)

ELIGIBILITY:
Inclusion Criteria:

* The patient has recurrent MDD, diagnosed according to DSM-5® and confirmed using the Mini-International Neuropsychiatric Interview (MINI).
* The patient has a MADRS total score ≥ 30 at the Screening Visit.
* As part of standard of care treatment, the patient is to be admitted to hospital due to the severity of the depressive symptoms and is willing to remain hospitalized for the duration of the study treatment period.
* The patient has had the current MDE for ≥3 months but less than 12 months.
* The patient has received treatment for the current episode with an SSRI/SNRI monotherapy (citalopram, escitalopram, paroxetine, duloxetine, venlafaxine, sertraline) at an approved dose for at least 6 weeks.

Exclusion criteria:

-The patient has any current psychiatric disorder or Axis I disorder (DSM-5® criteria), established as the primary diagnosis, other than MDD, as assessed using the MINI or another diagnostic interview

Other in- and exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day 0) to Day 1 (24 h post-infusion) in MADRS-6 subscale score | From baseline (Day 0) to Day 1 (24 h post-infusion)
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60. The primary endpoint will be evaluated with MADRS-6 subscale score, calculated based on the scores on MADRS items 1, 2, 3, 7, 8, and 9 which cover core symptoms (apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts) and is more sensitive to the effect of treatment.

SECONDARY OUTCOMES:
Change from baseline (Day 0) to Day 3 in MADRS-6 subscale score | From baseline (Day 0) to Day 3
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60. The endpoint will be evaluated with MADRS-6 subscale score, calculated based on the scores on MADRS items 1, 2, 3, 7, 8, and 9 which cover core symptoms (apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts) and is more sensitive to the effect of treatment.
Change from baseline (Day 0) to Day 7 in MADRS-6 subscale score | From baseline (Day 0) to Day 7
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60. The endpoint will be evaluated with MADRS-6 subscale score, calculated based on the scores on MADRS items 1, 2, 3, 7, 8, and 9 which cover core symptoms (apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts) and is more sensitive to the effect of treatment.
Change in MADRS total score from baseline to Day 1, Day 3, Day 7 | From baseline to Day 1, Day 3, Day 7
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60.
≥50% decrease in MADRS total score from baseline on Day 1 and Day 3 | On Day 1 and Day 3
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60.
CGI-I score at Day 1, Day 3, Day 7 | At Day 1, Day 3, Day 7
  The Clinical Global Impression (CGI) provides an overall clinician-determined summary measure that takes into account all available information, including knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI consists of two clinician-rated subscales: severity of illness (CGI-S) and global improvement (CGI-I). The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not.
CGI-I response (defined as CGI-I score ≤2) on Day 1 and 3 | At Day 1 and 3
  The Clinical Global Impression (CGI) provides an overall clinician-determined summary measure that takes into account all available information, including knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI consists of two clinician-rated subscales: severity of illness (CGI-S) and global improvement (CGI-I). The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not.
Change from baseline in CGI-S score to Day 1, Day 3, Day 7 | From baseline to Day 1, Day 3, Day 7
  The Clinical Global Impression (CGI) provides an overall clinician-determined summary measure that takes into account all available information, including knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI consists of two clinician-rated subscales: severity of illness (CGI-S) and global improvement (CGI-I). The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
CL/F of vortioxetine | Day 0, Day 1, Day 7
  Total plasma clearance of vortioxetine
Cav | Day 0, Day 1, Day 7
  average plasma concentration during a steady-state day

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (13):
- Bulgaria (8):
  - Mental Health Centre 'Prof. Dr. Ivan Temkov', EOOD (BG1004), Burgas
  - SPH - Kardzhali, EOOD (BG1005), Kardzhali
  - MHAT "Dr. Hristo Stambolski", EOOD (BG1001), Kazanlak
  - State Psychiatric Hospital "Sv. Ivan Rilski" (BG1009), Novi Iskar
  - UMHAT 'Dr. Georgi Stranski', EAD (BG1006), Pleven
  - MHC - Ruse, EOOD (BG1007), Rousse
  - State Psychiatric Hospital (BG1008), Tsarev Brod
  - Mental Health Center-Vratsa EOOD (BG1002), Vratsa
- Estonia (2):
  - Marienthali Kliinik (EE2001), Tallinn
  - Tartu University Hospital (EE2002), Tartu
- Latvia (3):
  - Psychoneurological Hospital of Daugavpils (LV3003), Daugavpils
  - Riga Centre of Psychiatry and Narcology (LV3002), Riga
  - Psychoneurological Hospital of Strenci (LV3001), Strenči

REFERENCES:
- [Derived] Rancans E, Zambori J, Dalsgaard M, Baayen C, Areberg J, Ettrup A, Florea I. Intravenous vortioxetine to accelerate onset of effect in major depressive disorder: a 7-day randomized, double-blind, placebo-controlled exploratory study. Int Clin Psychopharmacol. 2020 Nov;35(6):305-312. doi: 10.1097/YIC.0000000000000326. PMID 32784346